CLINICAL TRIAL: NCT04736979
Title: Antibiotic PRophylAxis Based on infeCTIve Risk in Cardiac Implantable Electronic Device - PRACTICE Study
Brief Title: Antibiotic PRophylAxis Based on infeCTIve Risk in Cardiac Implantable Electronic Device
Acronym: PRACTICE
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, Associate Professor, University Hospital of Ferrara
Other Study IDs: 170499
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Device Related Infection
Keywords: pacemaker; implantable cardioverter defibrillator; cardiac implantable electronic device; infection; antibiotic; Shariff score
MeSH Terms: conditions — Prosthesis-Related Infections; Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: amoxicillin clavulanate — dosage according to Shariff score and creatinine clearance

SUMMARY:
This study was aimed at the evaluation of a new protocol of antibiotic prophylaxis, stratified according to individual infective risk calculated with the Shariff score at the moment of cardiac implantable electronic device (CIED) implantation.

DETAILED DESCRIPTION:
Prospective, single centre, cohort study. Patients undergoing CIED surgery in a 3-years period were considered for participation. In particular, patients were eligible if undergoing first implantation or replacement or upgrade of pacemaker or implantable cardioverter-defibrillator (ICD), including cardiac resynchronization therapy (CRT).

At the time of enrolment, before index procedure, the Shariff score was calculated for every patient. According to the score, patients were stratified in two groups: low infective risk (score <3) and high infective risk (score ≥3). Two different protocols of antibiotic prophylaxis were administered according to risk stratification. Patients in the "low risk" group were treated with only two doses of antibiotics, both intravenous, of whom the first one hour before skin incision and the second after eight hours. Patients in the "high risk" group were treated with intravenous prophylaxis for two full days (of whom the first administration one hour before skin incision and the others every eight hours), followed by other seven days of oral prophylaxis, for a total of nine days. Thereby, every patient received one administration of intravenous antibiotic one hour before skin incision and a second administration after eight hours, while patients in the low risk group did not receive other antibiotics and patients in the high risk group continued intravenous antibiotics every eight hours for two days, followed by oral antibiotics for other seven days.

The intended drug for antibiotic prophylaxis was amoxicillin + clavulanic acid unless the patient had a history of allergic reactions to penicillin. The dosage was dependent on renal function: for intravenous amoxicillin + clavulanic acid 2.2 g in patients with creatinine clearance (CrCl) <30 ml/min and 1.2 g in patients with CrCl >30ml/min, for oral amoxicillin + clavulanic acid 1 g every 8 hours in patients with <30 ml/min and 1 g every 12 hours in patients with CrCl >30ml/min. In case of penicillin allergy, clindamycin was chosen. The intravenous dosage was 600 mg every 8 hours for CrCl <30 ml/min and 600 mg every 12 hours for CrCl >30 ml/min, while the oral dosage was 450 mg every 8 hours for CrCl <30 ml/min and 450 mg every 12 hours for CrCl >30 ml/min.

Patients who were already in antibiotic therapy at the time of index procedure (for reasons other than CIED implantation) were not stratified in one of the two groups: post-operative antibiotics were continued according to clinical indications and not to the study protocol. This group included patients with a documented or suspected infection before surgery in whom the CIED procedure was judged not deferrable.

ELIGIBILITY:
Inclusion Criteria:

* first implantation or replacement or upgrade of pacemaker or ICD

Exclusion Criteria:

* age 18 years
* ongoing pregnancy
* inability to express informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing CIED-related intervention
Sampling Method: Non-Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
CIED related infection | 6 months
  clinical diagnosis of systemic or local infection involving subcutaneous CIED pocket or intravenous/intracardiac CIED lead or sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, Principal Investigator — Università degli Studi di Ferrara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Malagu M, Vitali F, Brieda A, Cimaglia P, De Raffele M, Tazzari E, Musolino C, Balla C, Serenelli M, Cultrera R, Rapezzi C, Bertini M. Antibiotic prophylaxis based on individual infective risk stratification in cardiac implantable electronic device: the PRACTICE study. Europace. 2022 Mar 2;24(3):413-420. doi: 10.1093/europace/euab222. PMID 34487163